CLINICAL TRIAL: NCT01542177
Title: The Evaluation of Hypoxia Imaging in Patients With Pancreatic Cancer Using Positron Emission Tomography (PET) With 18F-Fluoroazomycin Arabinoside (18F-FAZA)
Brief Title: A Study Using 18F-FAZA and PET Scans to Study Hypoxia in Pancreatic Cancer
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Cancer Society (CCS) (Other)
Responsible Party: Sponsor
Other Study IDs: FAZA-Pancreas
Record Dates: First submitted 2012-01-05; First posted 2012-03-02 (Estimated); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Pancreatic Cancer; Hypoxia
Keywords: hypoxia; pancreas; cancer; pancreatic cancer; 18F-FAZA; 18F-Fluoroazomycin Arabinoside; Positron Emission Tomography; PET
MeSH Terms: conditions — Pancreatic Neoplasms; Hypoxia; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — 2 tubes of whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pancreatic cancer

SUMMARY:
This is a diagnostic study to look for low levels of oxygen (hypoxia) in pancreatic cancer using an imaging test called positron emission tomography (PET). Hypoxia can influence how pancreatic cancer grows and responds to treatments such as chemotherapy and radiotherapy. The use of PET scans to measure hypoxia may be better and simpler than the approaches used previously. This study will assess whether or not PET scans using a tracer called 18F-FAZA (18F-Fluoroazomycin Arabinoside) can provide useful information about hypoxia in pancreatic cancer. Also as part of the study, a blood sample will be taken to study biomarkers (substances in the body that may be important indicators of hypoxia and/or pancreatic cancer) that may be useful in studying pancreatic cancer and hypoxia.

DETAILED DESCRIPTION:
This is a single centre, single arm hypoxia study of pancreatic cancer with PET FAZA imaging.

PET-CT imaging of tumor hypoxia with FAZA will be done prior to the start of standard treatment for pancreatic cancer with chemotherapy. The FAZA PET-CT imaging session will last approximately 2.5 hours and include an initial dynamic scan to completely characterize the initial rapid phase of FAZA uptake, followed by a later static scan.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 18 years old
* Histologic diagnosis of pancreatic adenocarcinoma
* TNM (7th edition) cT1-4, N0-1, M0-1
* No cytotoxic anti-cancer therapy for advanced / metastatic pancreatic cancer prior to study entry
* Ability to provide written informed consent to participate in the study
* ECOG performance status 0, 1 or 2.
* Patient should have the following blood counts at baseline: ANC equal or greater to 1.5 x 109/L; Platelets equal or greater to 100 x 109/L; Hgb equal or greater to 9g/Dl
* Patient should have the following blood chemistry levels at baseline: AST (SGOT), ALT (SGPT) equal or less than 5 x upper limit of normal range (ULN) is allowed
* Patient has an identifiable tumor (pancreatic tumor and/or metastasis) by imaging (CT scan and/or MR)
* Patient must agree to use contraception considered adequate and appropriate by the investigator and if the patient is female of child-bearing potential, as evidenced by regular menstrual periods, she must have a negative serum pregnancy test (B-hCG)

Exclusion Criteria:

* Inability to lie supine for more than 30 minutes
* Any other type of primary cancer
* Life expectancy of less than 12 weeks
* Patient has known brain metastases unless previously treated and well controlled for at least 3 months (defined as stable clinically, no edema, no steroids and stable in two scans at least 4 weeks apart)
* Patient has serious medical risk factors involving any of the major organ systems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pancreatic cancer
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2012-02; Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Measure the hypoxia level in Patients with Pancreatic Cancer using Positron Emission Tomography (PET) with 18F-Fluoroazomycin Arabinoside (18F-FAZA). | 2 years

SECONDARY OUTCOMES:
Correlate FAZA PET uptake in pancreatic cancer with the extension of the disease. | 2 years
  Standardized uptake statistics will be calculated for each volume of interest (VOI): Maximum standardized uptake value (SUVMax), mean standardized uptake value (SUVMean) and standard deviation of standardized uptake values (SUVSD).
Correlate FAZA PET uptake in pancreatic cancer with CA 19-9 levels. | 2 years
  Standardized uptake statistics will be calculated for each volume of interest (VOI): Maximum standardized uptake value (SUVMax), mean standardized uptake value (SUVMean) and standard deviation of standardized uptake values (SUVSD). These parameters will be correlated with increasing or decreasing CA 19-9 levels (U/ml).
Correlate FAZA PET uptake in pancreatic cancer with tumor response. | 2 years
  Standardized uptake statistics will be calculated for each volume of interest (VOI): Maximum standardized uptake value (SUVMax), mean standardized uptake value (SUVMean) and standard deviation of standardized uptake values (SUVSD). Tumor response is measured in millimeters. Complete response is a tumor reduction of <5 mm, partial response is at least a 30% reduction, progressive disease is a 20% increase, and stable disease is no increase in shrinkage and no increase in growth.
Correlate FAZA PET uptake in pancreatic cancer with patient disease-free survival (DFS). | 2 years
  Kaplan-Meier actuarial method and/or the Cox proportional hazard model will be utilized.
Compare the pattern of FAZA uptake in different tumor sites (eg., lymph node metastases and liver metastasis). | 2 years
  Standardized uptake statistics will be calculated for each volume of interest (VOI): Maximum standardized uptake value (SUVMax), mean standardized uptake value (SUVMean) and standard deviation of standardized uptake values (SUVSD).
Determine the feasibility of using dynamic and static PET imaging of FAZA uptake in patients with pancreatic cancer. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: David Hedley, MD, Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada